CLINICAL TRIAL: NCT02466945
Title: Oral and Dental Tolerance and Efficacy on Dentinal Hypersensitivity of a Dental Gel, on Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DP30032015003
Record Dates: First submitted 2015-06-01; First posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-06

CONDITIONS: Dentinal Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- V063B-DP3003 (Other): all patients will received the study product (V063B-DP3003)
  Interventions: Device: V063B-DP3003

INTERVENTIONS:
Device: V063B-DP3003 — The medical device V063B-DP3003 has been developed to relieve and decrease dentinal hypersensitivity in patients by creating a film around the sensitive tooth in order to prevent pain. Application modalities: apply a pea size amount of product (around 0.5g) onto each of the sensitive teeth, 3 times a day, by gentle massage with clean finger after each brushing of teeth. Do not rinse

SUMMARY:
The aim of this clinical trial is to evaluate the tolerance and efficacy of a dental gel in patients with dentinal hypersensitivity.

DETAILED DESCRIPTION:
The aim of this clinical trial is to evaluate the tolerance and efficacy of dental gel V063B-DP3003 in patients with dentinal hypersensitivity, under normal conditions of use, under dentist control.

The primary objective of this study is to evaluate the global oral and dental tolerance of the studied product after 28 days of use.

Some efficacy objectives have been added to observe the efficacy of the dental gel. The dentinal hypersensitivity will be evaluated by the investigator with a thermal stimulus on two sensitive teeth selected by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged between18 and 70 years included
* Having signed his/her written informed consent,
* If it is a woman of childbearing potential :

Must have been using an effective method of contraception Negative Urine pregnancy test at inclusion,

* Subject who can be reached in case of emergency,
* Subject willing to be compliant to the protocol,
* Subject able to fill out the daily log and the questionnaire.
* Subject with at least 20 natural teeth (especially on the studied teeth),
* Subject with an healthy gum status according to the investigator,
* Subject with a mild to moderate dentinal hypersensitivity on at least 2 hypersensitive non adjacent teeth: with a Schiff cold air index from 1 to 2
* Subjects who show a response typical of sensitivity to the cold air blast at visit 1.

Exclusion Criteria:

* Subject participating to any other biomedical research projects,
* For women : Pregnant or breastfeeding,
* Has forfeited his/her freedom by administrative or legal award or is under guardianship,
* Subject who, in the judgement of the investigator, is not likely to be compliant during the study,
* Subject unable to understand the information given (for linguistic or psychiatric reasons) and to give his/her consent in writing,
* Subject having dental braces
* Subject having immune system disorder,
* Subject having asthma,
* Subject having a disease liable to interfere with study data according to the investigator,
* Subject with teeth showing evidence of facets of attrition, premature contact, cracked enamel on the tooth to be studied and adjacent teeth,
* Subject with teeth showing evidence of irreversible pulpitis and active periodontal disease,
* Subject having caries on the tooth to be studied and adjacent teeth
* Subject having restauration of any type in the tooth to be studied,
* Subject having occlusal overload or occlusal adjustment recently made in the tooth to be studied,
* Subject with crowns , bridges in the area of sensitivity,
* Subject had undergone professional desensitizing therapy during the 3 previous months,
* Subject having a cutaneous-mucosal disease liable to interfere with study data according to the investigator, especially: herpes or medical history herpes, aphtous and medical history of aphtous, lichen planus, chronic lupus erythematosis,
* Subject having undergone surgery, chemical or physical treatment to the concerned study area in the last 3 months,
* Subject allergic or intolerant to one of the components of the study product,
* Subject having a background of intolerance or allergy to cosmetics, drugs or to other substances (fruits, lactose intolerant, nuts, etc.),
* Subject planning to have any dental care during the study.
* Subject having a treatment liable to interfere with study data (aspirin or derivatives, anti-inflammatories, and other analgesic, antibiotics, antihistaminics, corticoids, desensitizing substances, immunosuppressants, calcic inhibitors and anticonvulsants) 2 days before the inclusion visit,
* Subject having used of over the counter product for dentinal hypersensitivity within the previous six weeks,
* Subject being vaccinated (4 weeks prior) or expecting to be vaccinated during the study,
* Subject having modified his/her cosmetic habits (on the areas concerned by the study) during the last 2 weeks,
* Subject having applied any local product the day of the inclusion visit on the study area except the usual toothpaste

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-03 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Global tolerance according to a 5-point grading scale taking into account physical signs observed and graded by the dentist and functionnal signs observed and graded by the patient | after 28 days
  The global tolerance of the product is assessed by the dentist after 28 days of use, rated on a 5-point grading scale(good tolerance, very good tolerance, good tolerance, moderate tolerance) . The results of the global tolerance will take into account the physical signs observed by the dentist and the functional signs observed by the patients during the study

SECONDARY OUTCOMES:
Cold air stimulus score on the schiff cold air index as a mesure of immediate efficacy | 5 and 60 minutes after application at day 1
  Immediate efficacy of the product at 5 and 60 minutes after application at day 1, according to Cold air Stimulus by delivered from a standard dental unit syringe and assessment of the score on the Schiff Cold air index with several measures.
Cold air stimulus score on the schiff cold air index as a mesure of short term efficacy | efficacy at day 4 and day 6
  Evaluate the short term efficacy of the product at Day 4 and Day 6, according to Cold air Stimulus by delivered from a standard dental unit syringe and assessment of the score on the Schiff Cold air index.
Cold air stimulus score on the schiff cold air index as a mesure of efficacy | between baseline and day 28
  Evaluate the efficacy on dentinal hypersensitivity of the product between baseline and day 28, according to Cold air Stimulus by delivered from a standard dental unit syringe and assessment of the score on the Schiff Cold air index.
Tolerance with the record of functionnal signs reported by the dentist and physical signs reported by the patient. | during 28 days
  Evaluate the oral and dental tolerance of the studied product thanks to functionnal signs reported and graded by the patient following a scale from 0=none to 4=severe and by the clinical examination of physical signs performed and graded by the investigator with a scale from 0=none to 4=severe
Acceptability of the product assessed with a questionnaire | during 28 days
  Evaluate acceptability with a questionnaire filled out by the subject on day 28.

OTHER OUTCOMES:
Safety of the product with the record of adverse event during the study | during 28 days
  collect Adverse events during the study

CONTACTS AND LOCATIONS:
Overall Officials: GARNER Kelly, Study Chair — Intertek Life Sciences; MACLURE Robert, MD, Principal Investigator — Intertek Life Sciences
Locations (1):
- Intertek Life Sciences, Cheshire, United Kingdom